CLINICAL TRIAL: NCT01465022
Title: Breastfeeding and Oral Contraceptives: a Randomized, Controlled Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of New Mexico (Other)
Collaborators: American College of Obstetricians and Gynecologists (Other)
Responsible Party: Principal Investigator, Eve Espey, Professor, OB-GYN, University of New Mexico
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 03-151
Record Dates: First submitted 2011-11-01; First posted 2011-11-04 (Estimated); Results first posted 2016-01-15 (Estimated); Last update posted 2016-05-20 (Estimated); Status verified 2016-02

CONDITIONS: Breast Feeding; Contraception
Keywords: Breastfeeding rates; Contraceptive continuation; Birth control pills; Lactation
MeSH Terms: conditions — Breast Feeding

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Study Arm A (Active Comparator): Study Arm A is one of two interventions (Combined estrogen-progestin pill)
  Interventions: Drug: Combined estrogen-progestin pill
- Study Arm B (Active Comparator): Study Arm B is one of two interventions (Progestin-only pill)
  Interventions: Drug: Progestin-only pill

INTERVENTIONS:
Drug: Combined estrogen-progestin pill — 1 mg norethindrone and .035 mg ethinyl estradiol orally for 21 days followed by 7 days of placebo
  Other Names: OCP
  Arms: Study Arm A
Drug: Progestin-only pill — .35 mg norethindrone once a day orally
  Other Names: POP
  Arms: Study Arm B

SUMMARY:
Objectives

To clarify the relationship between postpartum (2 weeks) use of progestin-only vs. combined oral contraceptive pills and the outcomes of breastfeeding continuation, infant growth, contraceptive method continuation, and pregnancy rates in breastfeeding women. Specific research questions:

1. To determine whether there is a difference in rates of breastfeeding continuation at 2 months and 4 months between postpartum breastfeeding women using progestin-only pills vs. combined pills.
2. To determine whether there is a difference in infant growth at 2 weeks and 8 weeks between postpartum breastfeeding women using progestin-only pills vs. combined pills.
3. To determine whether there is a difference in birth control method continuation at 2 months and 4 months between postpartum breastfeeding women using progestin-only pills vs. combined pills.

Hypothesis

Combined oral contraceptive pills, when initiated by postpartum breastfeeding women, will cause a differential in continuation of breastfeeding: 35% continuation in the combined pill group vs. 60% in the progestin-only pill group at 8 weeks.

ELIGIBILITY:
Inclusion Criteria:

* able to give informed consent
* postpartum women delivering at the University of New Mexico Hospital
* Intend to breastfeed
* Plan to use oral contraceptives as her family planning method
* Willing to be randomized to either progestin-only pills or combined pills

Exclusion Criteria:

* medical contraindications to combined pills including history of thromboembolism, uncontrolled hypertension or complex migraine headaches
* preterm birth (<37 weeks)
* small for gestational age infant (<2500 grams)
* large for gestational age infant (>4500 grams)
* infant with major congenital anomaly

Ages: 15 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 197 (Actual)
Dates: Start 2005-01; Primary Completion 2008-06 (Actual); Study Completion 2008-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Eve Espey, MD, Principal Investigator — UNM OB Gyn

REFERENCES:
- [Derived] Espey E, Ogburn T, Leeman L, Singh R, Ostrom K, Schrader R. Effect of progestin compared with combined oral contraceptive pills on lactation: a randomized controlled trial. Obstet Gynecol. 2012 Jan;119(1):5-13. doi: 10.1097/AOG.0b013e31823dc015. PMID 22143258

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study design is double-blind randomized controlled trial in which postpartum women who have decided to breastfeed and who choose birth control pills as their contraceptive method are randomized to one of two groups:
Pre-assignment Details: The research nurse recruiting the eligible subject will ask the subject if they have been given adequate time to make a decision regarding study participation.
Groups:
- Combined Estrogen-progestin Pill: Study Arm A is one of two interventions.
- Progestin-only Pill: Study Arm B is one of two interventions.
- Not Randomized: Participants who were consented but not randomized.
Period: Overall Study
Arm/Group | Combined Estrogen-progestin Pill | Progestin-only Pill | Not Randomized
Started | 64 | 63 | 70
Completed | 41 | 40 | 0
Not Completed | 23 | 23 | 70
Not completed — Lost to Follow-up | 15 | 14 | 0
Not completed — Breastfeeding discontinuation before 8 w | 8 | 9 | 0
Not completed — Not Randomized | 0 | 0 | 70

BASELINE CHARACTERISTICS:
Groups:
- Combined Estrogen-progestin Pill: Study Arm A is one of two interventions (OCP).
- Progestin-only Pill: Study Arm B is one of two interventions (POP).
- Not Randomized: 70 women who were enrolled.
- Total: Total of all reporting groups
Arm/Group | Combined Estrogen-progestin Pill | Progestin-only Pill | Not Randomized | Total
Number analyzed (Participants) | 64 | 63 | 70 | 197
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 64 | 63 | 70 | 197
  >=65 years | 0 | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 23.8 (4.4) | 25.0 (5.4) | 23.4 (5.0) | 24.4 (197)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 64 | 63 | 70 | 197
  Male | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 64 | 63 | 70 | 197

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Who Continued to Breastfeed at 6 Months
Description: Proportion of participants who are continuing to breastfeed from 2 months to 6 months after delivery
Time Frame: Baseline to Week 8, Week 8, 2-6 months
Population: Participants available for follow-up through a 6 month period
Measure: Number; unit: participants
Groups:
- Combined Estrogen-progestin Pill: Study Arm A is one of two interventions (Combined estrogen-progestin pill)
  Combined estrogen-progestin pill: 1 mg norethindrone and .035 mg ethinyl estradiol orally for 21 days followed by 7 days of placebo
- Progestin-only Pill: Study Arm B is one of two interventions (Progestin-only pill)
  Progestin-only pill: .35 mg norethindrone once a day orally
Arm/Group | Combined Estrogen-progestin Pill | Progestin-only Pill
Number analyzed (Participants) | 64 | 63
participants
  Particpants lost to follow-up | 15 | 14
  Discontinued Breastfeeding prior to 8 weeks | 8 | 9
  # of participants included in 8 week follow-up | 41 | 40
  Discontinued breastfeeding between 2-6 months | 13 | 14
  Participants available for follow-up at 6 months | 28 | 26

2. Secondary Outcome: Number of Participants Who Continued Birth Control Method After 6 Months
Description: Proportion of participants who are continuing to use either combined estrogen-progestin pill or progestin-only pill up to 6 months after delivery
Time Frame: Baseline to Week 8, Week 8, 2-6 months
Population: Participants available for follow-up through a 6 month period
Measure: Number; unit: participants
Arm/Group | Combined Estrogen-progestin Pill | Progestin-only Pill
Number analyzed (Participants) | 64 | 63
participants
  Particpants lost to follow-up | 15 | 14
  Discontinued oral contraceptives by 8 week mark | 1 | 0
  Participants available for follow-up at 8 weeks | 40 | 40
  Discontinued oral contraceptives from 2-6 months | 11 | 10
  Participants available for follow-up at 6 months | 29 | 30

3. Secondary Outcome: Infant Length Growth From 2-8 Weeks
Description: Comparison of infant length at 2 weeks and 8 weeks between postpartum breastfeeding women using progestin-only pills vs. combined pills. Inclusion criteria of mother's who are actively breastfeeding.
Time Frame: Week 2 and Week 8
Population: At 2 week point 64 participants for follow-up in combined pills arm, 63 for follow-up in progestin-only pills arm.
  At 8 week point 41 participants for follow-up in combined pills arm, 40 for follow-up in progestin-only pills arm.
Measure: Mean (Standard Deviation); unit: cm
Arm/Group | Combined Estrogen-progestin Pill | Progestin-only Pill
Number analyzed (Participants) | 64 | 63
cm
  Mean Infant length at 2 weeks | 51.5 (.49) | 51.7 (.49)
  Mean Infant length at 8 weeks | 56.8 (.49) | 57 (.49)

4. Secondary Outcome: Infant Weight Growth From 2-8 Weeks
Description: Comparison of infant growth at 2 weeks and 8 weeks between postpartum breastfeeding women using progestin-only pills vs. combined pills. Inclusion criteria of mother's who are actively breastfeeding.
Time Frame: Week 2 and Week 8
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: kg
Arm/Group | Combined Estrogen-progestin Pill | Progestin-only Pill
Number analyzed (Participants) | 64 | 63
kg
  Mean Infant weight at 2 weeks | 3.7 (.36) | 3.7 (.36)
  Mean infant weight at 8 weeks | 5.08 (.36) | 5.2 (.36)

5. Secondary Outcome: Infant Occipitofrontal Circumference Growth From 2-8 Weeks
Description: as for outcome 4
Time Frame: Week 2 and Week 8
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: cm
Arm/Group | Combined Estrogen-progestin Pill | Progestin-only Pill
Number analyzed (Participants) | 64 | 63
cm
  Infant occipitofrontal circumference at 2 weeks | 36 (.84) | 36.1 (.84)
  Infant occipitofrontal circumference at 8 weeks | 39 (.84) | 39 (.84)

ADVERSE EVENTS:
Time Frame: 3 years - no adverse events reported
Groups:
- Combined Estrogin-progestin Pill: Study Arm A is one of two interventions (Combined estrogen-progestin pill)
  Combined estrogen-progestin pill: 1 mg norethindrone and .035 mg ethinyl estradiol orally for 21 days followed by 7 days of placebo
Arm/Group | Combined Estrogin-progestin Pill | Progestin-only Pill
Serious Adverse Events (participants affected / at risk) | 0/64 | 0/63
Other Adverse Events (participants affected / at risk) | 0/64 | 0/63

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No